CLINICAL TRIAL: NCT06273969
Title: Protocol Development for Ultrasonographic Evaluation of the Effect of Osteopathic Manipulative Techniques on Thoracic Outlet Syndrome
Brief Title: Ultrasonographic Evaluation of Osteopathic Manipulation for Thoracic Outlet Syndrome
Acronym: TOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PK20240105-001
Record Dates: First submitted 2024-02-02; First posted 2024-02-23 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Thoracic Outlet Syndrome
Keywords: Blood Flow; Osteopathic Manipulation; Ultrasonography
MeSH Terms: conditions — Thoracic Outlet Syndrome | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Twelve consented male and/or female volunteers between the ages of 18 and 65 with intermittent tingling and/or numbness in one or both hands that has occurred with two weeks of the start date of the study will be evaluated using pulsed-wave doppler ultrasonography (US) and then treated with osteopathic manipulative treatment (OMT).
  US examination of the thoracic outlet will be performed using a Mindray-6 ultrasound machine and will include 4 views/positions with the subject in a seated position.
  The following intervention will consist of four osteopathic manipulation techniques (OMT) being performed that target the somatic dysfunctions associated with TOS. These techniques include: 1) Direct Thoracic Inlet Myofascial Release (TIMFR); 2) Direct Muscle Energy for the Scalene Muscles; 3) Direct Muscle Energy for the Pectoralis Muscles; and 4) Supraclavicular Fascial Release.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteopathic Manipulative Treatment (Experimental): The OMT protocol is designed to target the somatic dysfunction associated with TOS.
  Interventions: Other: Osteopathic Manipulative Treatment (OMT)

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment (OMT) — The OMT protocol is designed to target the somatic dysfunction associated with TOS. The somatic dysfunction associated with TOS include muscular hypertonicity of the anterior and middle scalene muscles, hypertonicity of the pectoralis muscles, and tension in the fascia of the supraclavicular area between the clavicle and first rib. The OMT protocol will consist of the following four techniques:
  Direct Thoracic Inlet Myofascial Release (TIMFR) - Reduce tension at the thoracic inlet fascia located between the thoracic outlet and the cervical spine.
  Direct Muscle Energy for the Scalene Muscles -Reduce tension within the scalene muscle group
  Direct Muscle Energy for the Pectoralis Muscles - Reduce tension within the pectoralis muscle group
  Supraclavicular Fascial Release - Reduce fascial tension within the supraclavicular fossa

SUMMARY:
The purpose of the study is to develop a protocol to assess blood flow in the upper limb vasculature before and after osteopathic manipulative treatment (OMT) using Pulsed-wave Doppler ultrasonography (US). We will assess the subclavian artery and vein at two locations (above and below the clavicle) and the brachial artery and vein (within the axilla) to determine the reproducibility of the blood flow findings at each location and the impact of OMT on the blood flow. Additionally we will qualitatively assess morphological changes of the brachial plexus before and after OMT with US.

DETAILED DESCRIPTION:
Thoracic outlet syndrome (TOS) includes a spectrum of symptoms caused by compression of neural or vascular structures in or near the superior thoracic aperture. TOS symptoms results when the subclavian vessels are obstructed or when the subclavian artery or vein, or brachial plexus are compressed by regional structures in or around the superior thoracic aperture causing numbness and tingling in the ipsilateral upper extremity.

OMT is a type of manual therapeutic approach used in the osteopathic profession that can be used to reduce symptoms in patients with TOS, but the underlying mechanisms of the treatment are unclear. Manual techniques, such as thoracic inlet myofascial release, can be used as part of a OMT approach to free local musculoskeletal restrictions around the brachial plexus and vasculature entering and exiting the upper extremity. The current evidence for the use of OMT in management of TOS is primarily limited to case studies.

More studies are required to determine whether OMT is effective and better understand why it might be effective. Currently, other treatments for TOS include physical therapy, trigger point injections, botulism injections, and acupuncture. Pharmacological treatments for TOS symptoms include muscle relaxants, antidepressants, anti-inflammatories such as NSAIDs and steroids, and anticoagulants-all of which have associated risks, contraindications, expenses, and side effects. Severe cases of TOS may require surgical decompression in the presence of severe symptoms that fail conservative treatments. OMT represents a quick conservative intervention that can be performed during an outpatient visit.

US is a noninvasive tool that can be used to evaluate blood flow in arteries and veins. In patients with TOS, US has shown significant changes in blood flow dynamics of the subclavian vessels. Significant changes were also seen in the subclavian artery blood flow during shoulder maneuvers (e.g. Adson's test, Wright's test, Elevated Arm Stress test, Roos test) that are used in the diagnostics of TOS. Therefore, it would be reasonable to use US to assess possible mechanisms by which OMT might reduce symptoms. Such information would allow physicians to understand how to use OMT techniques most effectively, either as an adjunct to other treatments, or as standalone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years of age
* Experienced intermittent tingling and/or numbness in one or both hands that has occurred within two weeks of the start date of this study.

Exclusion Criteria:

* Pregnant
* Body mass index (BMI) over 30 kg/m2 (obese)
* Prior surgery, broken bones, or known birth defects affecting the thoracic outlet, such as clavicular fracture or congenital first rib

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Blood flow changes in the upper extremity. | Pre and post osteopathic manipulative treatment on the day of treatment. Pre-measurement followed by 10 minutes of rest before OMT. Post-measurement made immediately following the OMT treatment.
  Changes in blood flow to the upper extremity in participants who have been experiencing TOS symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kondrashov, PhD, Principal Investigator — A.T. Still University
Locations (1):
- A.T. Still University, Kirksville, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen H, Baker N, Williams K, Criado E. Physiologic variations in venous and arterial hemodynamics in response to postural changes at the thoracic outlet in normal volunteers. Ann Vasc Surg. 2014 Oct;28(7):1583-8. doi: 10.1016/j.avsg.2014.05.003. Epub 2014 Jun 6. PMID 24909503
- [Background] Cocco G, Ricci V, Ricci C, Nanka O, Catalano O, Corvino A, Boccatonda A, Serafini FL, Izzi J, Vallone G, Cantisani V, Iannetti G, Caulo M, Ucciferri C, Vecchiet J, Pizzi AD. Ultrasound imaging of the axilla. Insights Imaging. 2023 May 11;14(1):78. doi: 10.1186/s13244-023-01430-9. PMID 37166516
- [Background] Kimberly PE, Halma K. Outline of osteopathic manipulative procedures: the Kimberly manual 2006. Marceline (MO): Walsworth Publishing; 2008.
- [Background] Kuchera ML, Wallace E. Lymphatic drainage procedures. In: Seffinger MA, editor. Foundations of osteopathic medicine: philosophy, science, clinical applications, and research. 4th ed. Philadelphia (PA): Wolters Kluwer; 2018. p. 906-922.
- [Background] Dalley AF 2nd, Agur AMR. Moore's clinically oriented anatomy. 9th ed. Philadelphia (PA); Wolters Kluwer; 2023.
- [Background] Nicholas AS, Nocholas EA. Atlas of osteopathic techniques. 4th ed. Philadelphia (PA): Wolters Kluwer; 2023.
- [Background] Hussain MA, Aljabri B, Al-Omran M. Vascular Thoracic Outlet Syndrome. Semin Thorac Cardiovasc Surg. 2016 Spring;28(1):151-7. doi: 10.1053/j.semtcvs.2015.10.008. Epub 2015 Oct 28. PMID 27568153
- [Background] Huang JH, Zager EL. Thoracic outlet syndrome. Neurosurgery. 2004 Oct;55(4):897-902; discussion 902-3. doi: 10.1227/01.neu.0000137333.04342.4d. PMID 15458598
- [Background] Lapegue F, Faruch-Bilfeld M, Demondion X, Apredoaei C, Bayol MA, Artico H, Chiavassa-Gandois H, Railhac JJ, Sans N. Ultrasonography of the brachial plexus, normal appearance and practical applications. Diagn Interv Imaging. 2014 Mar;95(3):259-75. doi: 10.1016/j.diii.2014.01.020. Epub 2014 Mar 3. PMID 24603038
- [Background] Moore R, Wei Lum Y. Venous thoracic outlet syndrome. Vasc Med. 2015 Apr;20(2):182-9. doi: 10.1177/1358863X14568704. PMID 25832605
- [Background] Pisko-Dubienski ZA, Hollingsworth J. Clinical application of Doppler ultrasonography in the thoracic outlet syndrome. Can J Surg. 1978 Mar;21(2):145-7, 150. PMID 630465
- [Background] Stapleton C, Herrington L, George K. Sonographic evaluation of the subclavian artery during thoracic outlet syndrome shoulder manoeuvres. Man Ther. 2009 Feb;14(1):19-27. doi: 10.1016/j.math.2007.07.010. Epub 2007 Oct 24. PMID 17928256
- [Background] Sucher BM. Ultrasonography-guided osteopathic manipulative treatment for a patient with thoracic outlet syndrome. J Am Osteopath Assoc. 2011 Sep;111(9):543-7. doi: 10.7556/jaoa.2011.111.9.543. PMID 21955534
- [Background] Vemuri C, McLaughlin LN, Abuirqeba AA, Thompson RW. Clinical presentation and management of arterial thoracic outlet syndrome. J Vasc Surg. 2017 May;65(5):1429-1439. doi: 10.1016/j.jvs.2016.11.039. Epub 2017 Feb 8. PMID 28189360
- [Background] Wadhwani R, Chaubal N, Sukthankar R, Shroff M, Agarwala S. Color Doppler and duplex sonography in 5 patients with thoracic outlet syndrome. J Ultrasound Med. 2001 Jul;20(7):795-801. doi: 10.7863/jum.2001.20.7.795. PMID 11444739
- [Background] Yuschak E, Haq F, Chase S. A Case of Venous Thoracic Outlet Syndrome: Primary Care Review of Physical Exam Provocative Tests and Osteopathic Manipulative Technique Considerations. Cureus. 2019 Jun 17;11(6):e4921. doi: 10.7759/cureus.4921. PMID 31423397
- [Background] Cavanna AC, Giovanis A, Daley A, Feminella R, Chipman R, Onyeukwu V. Thoracic outlet syndrome: a review for the primary care provider. J Osteopath Med. 2022 Aug 29;122(11):587-599. doi: 10.1515/jom-2021-0276. eCollection 2022 Nov 1. PMID 36018621
- [Background] Jones MR, Prabhakar A, Viswanath O, Urits I, Green JB, Kendrick JB, Brunk AJ, Eng MR, Orhurhu V, Cornett EM, Kaye AD. Thoracic Outlet Syndrome: A Comprehensive Review of Pathophysiology, Diagnosis, and Treatment. Pain Ther. 2019 Jun;8(1):5-18. doi: 10.1007/s40122-019-0124-2. Epub 2019 Apr 29. PMID 31037504
- [Background] Kim M, Chi EH, Lee J, Ha I. The clinical observation of muscle energy techniques of ligamentous articular strain in 2 cases of cervical disc herniation with thoracic outlet syndrome. Int J of Osteo Med. 2015; 18: 63-70.